CLINICAL TRIAL: NCT02677961
Title: An Electronic Health Record (EHR)-Based Comprehensive Bone and Soft Tissue Tumor Registry
Status: Recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, David Liebner, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-14242
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Neoplasms, Connective and Soft Tissue; Bone Neoplasms
Keywords: sarcoma; registry
MeSH Terms: conditions — Neoplasms, Connective and Soft Tissue; Bone Neoplasms; Sarcoma | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation

SUMMARY:
Translational studies in cancer research can be impeded by the lack of high-quality clinical data that can be correlated with research questions. This is particularly true in the case of rare diseases, such as bone and soft tissue tumors. It is therefore the purpose of this study to create a prospective EHR-based clinical registry for individuals with bone and soft-tissue tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To create a secure EHR-based registry to allow for the prospective collection of clinical and research data in a collection of rare diseases (bone and soft-tissue tumors).

II. To facilitate the identification and validation of clinical and molecular features that may be associated with prognosis and/or response to therapy in (subtypes) of bone and soft-tissue tumors.

III. To pilot a mechanism that will facilitate future collaboration between institutions for research and analysis of bone and soft-tissue tumors.

IV. To standardize biospecimen collection for correlative biomarker analysis for patients undergoing treatment and surveillance for bone and soft tissue tumors at Ohio State University.

OUTLINE: This is an observational study.

Patients complete quality of life questionnaires and their medical records are reviewed. Patients may also undergo collection of blood samples for up to 2 years, unless otherwise specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis or presumed diagnosis of bone or soft tissue tumor as defined by the WHO classification of tumors of soft tissue and bone (4th ed.)
* Patient, or his/her designated power of attorney, must be able to understand and approve of the consent to participate.

Exclusion Criteria:

* Prisoners are excluded from participation in the Registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of bone or soft-tissue tumor as defined by the WHO classification of tumors of soft tissue and bone (4th ed.)
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: David A Liebner, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu